CLINICAL TRIAL: NCT00824941
Title: Brain-Gut Interactions in Overweight and Normal Weight Patients With Chronic Abdominal Pain
Status: Terminated | Type: Observational
Sponsor: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 090064; 09-NR-0064
Record Dates: First submitted 2009-01-16; First posted 2009-01-19 (Estimated); Last update posted 2019-11-20 (Actual); Status verified 2019-11-13

CONDITIONS: Obesity; Stress; Irritable Bowel Syndrome; Women; Abdominal Pain
Keywords: Abdominal Pain; Women's Health and Disease; Inflammation; Symptoms; Brain; Chronic Abdominal Pain
MeSH Terms: conditions — Obesity; Irritable Bowel Syndrome; Abdominal Pain; Disease; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

SUMMARY:
About 15 to 20 percent of individuals living in the United States have chronic abdominal pain, often of unknown origin, which is often difficult to diagnose and treat. One possible cause of chronic abdominal pain is an inflammation of the intestines, but it is not known whether the two are related. Furthermore, although overweight people tend to be more likely to have increased inflammation, it is not known whether there is a connection between increased body weight and chronic abdominal pain. This study will examine the relationship between symptoms of chronic abdominal pain and intestinal inflammation by comparing the medical test results of normal weight and overweight patients who have a history of chronic abdominal pain.

This study will include 224 subjects, who must be men and women between the ages of 13 and 45. Half the subjects will be healthy participants, and half will have had chronic abdominal pain of unknown origin for longer than 6 months. Female participants must take a urine pregnancy test before starting the study, and will not be allowed to participate if the test is positive. During the study, patients will visit the NIH Clinical Center on two occasions for testing.

On the first visit, patients will provide a medical history, including information about current medications or natural remedies and tobacco and alcohol use, and will also fill out questionnaires to provide information about symptoms, current levels of gastrointestinal pain, and general quality of life. The study researchers will conduct a physical examination, measure patients height and weight, and draw blood for testing.

Patients will be asked to not eat or drink anything for 8 hours before the second visit, and will be asked to bring a bathing suit and a swim cap to the Clinical Center. On the day of the visit, patients will fill out questionnaires to provide information about symptoms, current levels of gastrointestinal pain, and general quality of life. Patients will also provide a blood sample for testing. Researchers will measure patients blood pressure and heart rate, height, weight, waist/hip circumference, and intra-abdominal measurement. Patients will also be asked to put on the bathing suit and swim cap to have their body fat measured using a machine called the BOD POD. To test the gastrointestinal system, patients will then be asked to drink a sugar-based test solution, and researchers will collect all voided urine for the next 5 to 6 hours. (Patients may drink water during this time.)

On either Day 1 or Day 2 of the study, patients will sip, swish and spit an additional sweet taste solution. Patients will sip, swish, and spit different concentrations of this sweet taste solution, for a total of 25 tastings of this solution. Subjects will then complete questionnaires about their sweetness preferences related to these 25 tastings.

DETAILED DESCRIPTION:
The objective of this natural history study is to assess the specific gastrointestinal (GI) symptoms and pathophysiology of chronic abdominal pain of unknown origin at the molecular level. This research will test the hypothesis that chronic abdominal pain of unknown etiology has an inflammatory mechanism. Although increased body weight may be associated with increased inflammation, it is unclear that increased body weight is associated with chronic abdominal pain. Accordingly both overweight and normal weight subjects with and without chronic abdominal pain of unknown origin will be included in this study. The study design is a longitudinal natural history.

The purpose is to test the relationship between abdominal pain symptoms and intestinal inflammation in two groups (overweight and normal weight patients with chronic abdominal pain of unknown origin). After obtaining informed consent, an initial screening history and physical exam to ensure eligibility will be performed. The participants abdominal pain, psychological distress, quality of life, socio-demographic, and co-morbidities will be assessed via questionnaires. Anthropometry, vital signs, and fasting blood work will be drawn at both of the two visits to the Clinical Center of the National Institutes of Health for clinical screening labs and research purposes.

There are three measures of intestinal inflammation including fecal calprotectin, intestinal permeability, and serum cytokine IL-6 levels. A stool sample will be collected to measure fecal calprotectin. Intestinal permeability will be measured with the administration of a sugar based test solution which will be given orally to participants after an overnight fast on their second visit. Excreted urine sugar ratios, expressed per m2 of body surface area, will measure gastrointestinal permeability. Body mass and body fat analysis (plethysmography), intra-abdominal and liver ultrasound, and Fibroscan measures will also be collected on visit two. On either Day 1 or Day 2 of the study, patients will sip, swish and spit additional sweet taste solutions and complete questionnaires about their sweetness preferences related to these tastings.

ELIGIBILITY:
* INCLUSION CRITERIA:

To be included, patients must meet all of the following:

* Have a history of abdominal pain for greater than 6 months
* Males ages 13-45 years old or females ages 13-45 years old who have had their menses for at least 2 years
* Provide written informed consent, prior to entering the study or undergoing any study procedures

EXCLUSION CRITERIA:

Patients with any of the following will be excluded:

* Have a history of an organic GI disease (e.g., inflammatory bowel disease, celiac disease, biliary disorders, bowel resection) cardiac, pulmonary, neurologic, renal, endocrine, or gynecological pathology
* Are currently taking medications for GI symptoms daily such as 5-HT3 antagonists/5-HT4 agonists, prokinetic drugs, laxatives (but not fiber supplements), anti-diarrheals or antispasmodics
* Are currently taking other medications daily that would alter serotonin (e.g., serotonin specific reuptake inhibitors [SSRI]), catecholamines (e.g., tricycle antidepressants but not inhaled beta-agonist for mild-moderate asthma), cortisol (excluding inhaled corticosteroids)
* Work during the late evening and night (as cortisol levels may be altered)
* Severe co-morbid pain or psychiatric conditions (e.g., fibromyalgia, bipolar or psychotic disorder)
* Take greater than 300 mg of caffeine containing beverages or food (e.g. chocolate) in the afternoon-evening or greater than 2 servings of alcohol containing beverages everyday (decaffeinated coffee is acceptable)
* Are unable to give informed consent
* Are unable to physically use the touch screen for the purpose of the study
* Are visually impaired or currently institutionalized
* Females who are pregnant or lactating
* NINR employees, subordinates/relatives/ or co-workers
* Any NIH employee who is a subordinate/relative/or co-worker of a study investigator

Ages: 13 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 132 (Actual)
Dates: Start 2009-02-06; Study Completion 2019-11-13

PRIMARY OUTCOMES:
No intervention. Natural history study | At enrollment
  Compare abdominal pain and intestinal inflammation in normal weight and overweight individuals.

SECONDARY OUTCOMES:
Natural History study. | At enrollment
  Characterize association between abdominal pain and inflammatory markers.

CONTACTS AND LOCATIONS:
Overall Officials: Wendy A Henderson, C.R.N.P., Principal Investigator — National Institute of Nursing Research (NINR)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Creed F, Ratcliffe J, Fernandez L, Tomenson B, Palmer S, Rigby C, Guthrie E, Read N, Thompson D. Health-related quality of life and health care costs in severe, refractory irritable bowel syndrome. Ann Intern Med. 2001 May 1;134(9 Pt 2):860-8. doi: 10.7326/0003-4819-134-9_part_2-200105011-00010. PMID 11346322
- [Background] Russo MW, Gaynes BN, Drossman DA. A national survey of practice patterns of gastroenterologists with comparison to the past two decades. J Clin Gastroenterol. 1999 Dec;29(4):339-43. doi: 10.1097/00004836-199912000-00009. PMID 10599638
- [Background] Mayer EA. The neurobiology of stress and gastrointestinal disease. Gut. 2000 Dec;47(6):861-9. doi: 10.1136/gut.47.6.861. No abstract available. PMID 11076888
- [Derived] Joseph PV, Davidson HR, Boulineaux CM, Fourie NH, Franks AT, Abey SK, Henderson WA. Eating Behavior, Stress, and Adiposity: Discordance Between Perception and Physiology. Biol Res Nurs. 2018 Oct;20(5):531-540. doi: 10.1177/1099800418779460. Epub 2018 May 31. PMID 29852756
- [Derived] Abey SK, Yuana Y, Joseph PV, Kenea ND, Fourie NH, Sherwin LB, Gonye GE, Smyser PA, Stempinski ES, Boulineaux CM, Weaver KR, Bleck CK, Henderson WA. Lysozyme association with circulating RNA, extracellular vesicles, and chronic stress. BBA Clin. 2016 Dec 20;7:23-35. doi: 10.1016/j.bbacli.2016.12.003. eCollection 2017 Jun. PMID 28053879
- [Derived] Del Valle-Pinero AY, Sherwin LB, Anderson EM, Caudle RM, Henderson WA. Altered vasoactive intestinal peptides expression in irritable bowel syndrome patients and rats with trinitrobenzene sulfonic acid-induced colitis. World J Gastroenterol. 2015 Jan 7;21(1):155-63. doi: 10.3748/wjg.v21.i1.155. PMID 25574088
- [Derived] Reddy SY, Rasmussen NA, Fourie NH, Berger RS, Martino AC, Gill J, Longchamps R, Wang XM, Heitkemper MM, Henderson WA. Sleep quality, BDNF genotype and gene expression in individuals with chronic abdominal pain. BMC Med Genomics. 2014 Oct 31;7:61. doi: 10.1186/s12920-014-0061-1. PMID 25358868
- [Derived] Del Valle-Pinero AY, Martino AC, Taylor TJ, Majors BL, Patel NS, Heitkemper MM, Henderson WA. Pro-inflammatory chemokine C-C motif ligand 16 (CCL-16) dysregulation in irritable bowel syndrome (IBS): a pilot study. Neurogastroenterol Motil. 2011 Dec;23(12):1092-7. doi: 10.1111/j.1365-2982.2011.01792.x. Epub 2011 Sep 23. PMID 21951809